CLINICAL TRIAL: NCT03370185
Title: A Phase 2 Study of Duvelisib Efficacy and Safety in Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) Previously Treated With a Bruton's Tyrosine Kinase Inhibitor (BTKi)
Brief Title: Phase 2 Study of Duvelisib in Previously Treated Patients With Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma
Acronym: BRIO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Reassessing corporate priorities.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-0145-224
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Leukemia; Lymphoma; Refractory; Relapse
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma; Recurrence | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib (Experimental): Duvelisib 25 mg orally (PO) twice daily (BID) continuously in 28-day cycles
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Duvelisib 25 mg orally (PO) twice daily (BID) continuously in 28-day cycles

SUMMARY:
This is a multi-center, single-arm, open-label, Phase 2 study of duvelisib, an orally bioavailable dual inhibitor of PI3K-δ,γ, in patients with CLL/SLL who have previously been treated with ibrutinib or another Bruton's Tyrosine Kinase Inhibitor (BTKi) and relapsed or were refractory to such therapy or discontinued such therapy due to toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Diagnosis of CLL or SLL.
3. Received at least one prior anti-cancer therapy for CLL or SLL.
4. Previous exposure to BTKi and meet at least one of the criteria below:

   1. Progressive disease (PD) while receiving or within 6 months after completing BTKi therapy.
   2. Discontinued a BTKi therapy due to BTKi treatment- related intolerance.
5. Measurable disease with a lymph node or tumor mass > 1.5 cm in at least one dimension.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Resolution of toxicities due to prior BTKi therapy to acceptable level.
8. Willingness of male and female patients to use medically acceptable methods of birth control.
9. Willing and able to participate in all required study evaluations and procedures.

Exclusion Criteria:

1. Richter's transformation or prolymphocytic leukemia
2. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
3. Received prior transplant
4. Experienced PD or serious adverse events on a prior phosphoinositide-3-kinase (PI3K) inhibitor
5. Known central nervous system involvement by CLL/SLL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From start of treatment to first documented response, 2 cycles (58 days)

SECONDARY OUTCOMES:
Treatment-Emergent adverse events (TEAEs) and changes in laboratory values | From start of treatment to end of treatment plus 30 days; 7 months
Duration of response (DOR), defined as the time from the first documentation of response to the first documentation of PD or death due to any cause | Time from the first documentation of response to first documentation of progressive disease or death due to any cause, 6 months
Progression-free survival (PFS), defined as the time from the first dose of study treatment to the first documentation of PD or death from any cause | Time from start of treatment to first documentation of progression or date of death from any cause, whichever came first, 4 months
Disease control rate (DCR), defined as CR/CRi + PR/PRwL + stable disease (SD) ≥ 8 weeks | Greater than or equal to 8 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Oncology, Tempe, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Ingalls Memorial Hospital, Harvey, Illinois
  - QUEST Research Institute, Royal Oak, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Summit Medical Group, Morristown, New Jersey
  - Medical Oncology Associates PS, WA, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No